CLINICAL TRIAL: NCT00594438
Title: Randomized, Prospective Comparison of Two Femoral Reaming Systems
Acronym: RIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Synthes Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F061204007
Record Dates: First submitted 2007-12-21; First posted 2008-01-15 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Femur Fracture
Keywords: Synthes Reamer-Irrigator-Aspirator (RIA); Zimmer Sentinal Reamer; Transesophageal Echocardiogram (TEE)
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1, A (Experimental): Femoral reaming with the Synthes Reamer-Irrigator-Aspirator (RIA)
  Interventions: Device: Synthes Reamer-Irrigator-Aspirator (RIA)
- 2 B (Active Comparator): Femoral reaming with a Zimmer Sentinel Reamer.
  Interventions: Device: Zimmer Sentinel Reamer

INTERVENTIONS:
Device: Synthes Reamer-Irrigator-Aspirator (RIA) — A standard lateral approach to the proximal femur will be utilized. The starting point will be identified using a guide pin and fluoroscopy using standard technique. The attending surgeon will perform the case from the opening of the canal with a drill through the completion of reaming. A transesophageal echocardiogram (TEE) will be recorded from the time the initial reamer engages the cortex until it is removed from the bone. A guide wire will be passed across the fracture site and its position confirmed by fluoroscopic imaging. The femoral canal will be reamed using the RIA device.
  Other Names: Reamer-Irrigator-Aspirator, Synthes
  Arms: 1, A
Device: Zimmer Sentinel Reamer — A standard lateral approach to the proximal femur will be utilized. The starting point will be identified using a guide pin and fluoroscopy using standard technique. The attending surgeon will perform the case from the opening of the canal with a drill through the completion of reaming. A transesophageal echocardiogram TEE will be recorded from the time the initial reamer engages the cortex until it is removed from the bone. A guide wire will be passed across the fracture site and its position confirmed by fluoroscopic imaging. The femoral canal will be reamed using either a conventional reaming technique or the RIA device.
  Arms: 2 B

SUMMARY:
The purpose of this study is to compare the quantity of fat that is released into the venous system (blood) by reaming the femoral canal during intramedullary nailing of the femur using two different reaming systems.

DETAILED DESCRIPTION:
Twenty patients who meet criteria for inclusion in this study will be assigned to one of two groups by means of a computer-generated random number. Group A will consist of 10 patients who undergo reaming with the Synthes reamer-irrigator-aspirator (RIA). Group B will consist of 10 patients who undergo conventional reaming with the Zimmer Sentinel reamer.

The patient will be transported to the operating room and will undergo general anesthesia. After correct positioning of the patient on the radiolucent table, baseline data will be collected. This data will consist of a transesophageal echocardiogram (TEE) and arterial blood gas.

A standard lateral approach to the proximal femur will be utilized. The starting point will be identified using a guide pin and fluoroscopy using standard technique. Though the resident may perform the approach, the attending surgeon will perform the case from the opening of the canal with a drill through the completion of reaming. A TEE will be recorded from the time the initial reamer engages the cortex until it is removed from the bone. A guide wire will be passed across the fracture site and its position confirmed by fluoroscopic imaging. The femoral canal will be reamed using either a conventional reaming technique or the RIA device.

For conventional reaming, successive reamers will be used beginning with an 8mm end-cutting reamer and increasing by 1.0 mm increments until cortical "chatter" is detected, then reaming will proceed at 0.5 mm increments for two passes. This is the standard practice using current technology. A Synthes titanium nail of the appropriate length which is 1.0 - 1.5mm less than the last reaming will be chosen for implantation. TEE will be monitored during the pass of the first reamer and the last.

For reaming with the RIA, a reamer-irrigator-aspirator of the appropriate size based on pre-operative evaluation of the femoral canal size will be used to perform a single pass down the femoral canal. A Synthes titanium femoral nail of the appropriate length will be selected for implantation. TEE will be recorded during the reaming. An arterial blood gas will be sent after positioning of the patient, when the guide wire is passed down the femoral canal and after the proximal locking screws are placed.

Proximal and distal locking screws will be placed in standard fashion. Wound closure and post-operative care will be according to standard protocols.

The TEE will be evaluated in a blinded manner by two anesthesiology attendings certified to use and evaluate the TEE. A grading system of 1 through 5 will be used, with 1 representing little to no fat emboli and 5 representative of a large number of fat emboli. This data will be forwarded to the principal investigator and used to fill the appropriate data sheet.

Outpatient follow-up will be performed in the usual manner, with sutures/staples being removed at approximately 2 weeks, and radiographs being obtained at 6 and 12 weeks as the attending physician deems clinically necessary. Follow-up for both limbs of the study will be the same as patients not in the study who undergo femoral nailing.

ELIGIBILITY:
Inclusion Criteria:

* injuries include isolated or multiple trauma which includes a femur fracture requiring operative fixation using an intramedullary nail using antegrade approach
* Adult patients ages 19-50 years old

Exclusion Criteria:

* pathologic fractures
* femoral deformities which would preclude intramedullary nailing
* pregnancy
* previous ipsilateral femoral nailing
* pediatric femoral fractures (<19 years old)

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Determine which of 2 femoral reamers is best for patients. | Surgery: 2-3 hours; Follow-up: 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: David A Volgas, MD, Principal Investigator — The University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Orthopaedic Trauma, Birmingham, Alabama, United States